CLINICAL TRIAL: NCT06655571
Title: What Technique for Caudal Block in Children: Conventional or Ultrasound-guided
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Mehdi Trifa, Head of the anesthesia and intensive care department, Tunis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 172024
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Compare Ultrasound-guided Caudal Block to the Conventional Technique Based on Anatomical Landmarks
Keywords: caudal block - children - ultrasound - conventional method

STUDY DESIGN:
Intervention Model Description: caudal block based on anatomical landmarks (group C) or ultrasound-guided (group E)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ultrasound (Other): Caudal bloc guided by Ultrasound
  Interventions: Procedure: Ultrasound guided caudal Block
- Conventionel (Other): Caudal Block based on anatomical landmarks
  Interventions: Procedure: Conventionel

INTERVENTIONS:
Procedure: Ultrasound guided caudal Block — caudal block using Ultrasound
  Arms: ultrasound
Procedure: Conventionel — Caudal Block based on anatomical landmarks
  Arms: Conventionel

SUMMARY:
The goal of our study is to compare ultrasound-guided caudal block to the conventional technique based on anatomical landmarks.

DETAILED DESCRIPTION:
The primary endpoint was the success rate of each technique. We also collected the time taken for each technique, the number of punctures, and the incidence of complications (subcutaneous infiltration, intravascular injection).

Children were randomized to receive a caudal block based on anatomical landmarks (group C) or ultrasound-guided (group E) at a dose of 1 ml/kg of 0.25% bupivacaine, not exceeding 20 ml.

ELIGIBILITY:
Inclusion Criteria:

* children aged between 6 months and 6 years, ASA 1 , underwent elective surgery

Exclusion Criteria:

* severe systemic diseases, previous neurological or spinal disorders, coagulation abnormalities, allergies toward LAs, local infection at the block site

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of block | during surgery
  A successful block was defined as an absence of significant motor movements following surgical induction or aberrations in the heart or respiratory rates

SECONDARY OUTCOMES:
block performing time | perioperative
  the period between anatomical structures identification and termination of LA administration
number of needle puncture | during procedure
complication rates | during procedure
  Blood aspiration Subcutaneous bulging Bone contact Dural puncture Local anesthetic toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Bechir Hamza hospital, Tunis, Tunis Governorate, Tunisia